CLINICAL TRIAL: NCT02385539
Title: Intrathecal Anesthesia for Elderly Patients Undergoing Surgery Lasting >45 Minutes: A Randomized, Controlled, Dose and Combination Finding Study
Brief Title: Intrathecal Administration of Levobupivacaine and Opioids in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Šarić, Jadranka Pavičić, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JPAVSAR
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Adverse Reaction to Spinal Anesthetic
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levobupivacaine (LB) 6 mg (Active Comparator): Patients will be stratified into three groups (80 patients) according to doses of Levobupivacaine (6, 8 or 12 mg, Chirocaine, Abbot Laboratories, amp. 5 mg/ml). Patients who will receive 6 mg of Levobupivacaine will be randomized to one of four treatment groups (each 20 patients), by dose of intrathecal opioids: 25, 35 mcg of Fentanyl (Fentanyl, Janssen Cilag, amp. 50 mcg/ml) or 5, 7 mcg of Sufentanil (Sufenta, Janssen-Pharmaceutica, amp. 5 mcg/ml). The groups will be named according to dose and combination of Levobupivacaine and Fentanyl or Sufentanil that will be given intrathecally as LB6F25 (LB 6 mg, Fentanyl 25 mcg), LB6F35 (LB 6 mg, Fentanyl 35 mcg), LB6S5 (LB 6 mg, Sufentanil 5 mcg), LB6S7 (LB 6 mg, Sufentanil 7 mcg). Hemodynamic and opioid's side effects will be recorded. The level and duration of sensory block, time until two-segment regression, T12 regression andl full skin sensory sensibility at the S1 segment will be registered
  Interventions: Drug: The impact of 10 independent variables on the likelihood of not developing hypotension after intrathecal injection.
- Levobupivacaine (LB) 8 mg (Active Comparator): Patients will be stratified into three groups (80 patients) according to doses of Levobupivacaine (6, 8 or 12 mg, Chirocaine, Abbot Laboratories, amp. 5 mg/ml). Patients who will receive 8 mg of Levobupivacaine will be randomized to one of four treatment groups (each 20 patients), by dose of intrathecal opioids: 25, 35 mcg of Fentanyl (Fentanyl, Janssen Cilag, amp. 50 mcg/ml) or 5, 7 mcg of Sufentanil (Sufenta, Janssen-Pharmaceutica, amp. 5 mcg/ml). The groups will be named according to dose and combination of Levobupivacaine and Fentanyl or Sufentanil that will be given intrathecally as LB8F25 (LB 8 mg, Fentanyl 25 mcg), LB8F35 (LB 8 mg, Fentanyl 35 mcg), LB8S5 (LB 8 mg, Sufentanil 5 mcg), LB8S7 (LB 8 mg, Sufentanil 7 mcg). Hemodynamic and opioid's side effects will be recorded after intrathecal injection. The level and duration of sensory block, time until two-segment regression, T12 regression andl full skin sensory sensibility at the S1 segment will be registered
  Interventions: Drug: The impact of 10 independent variables on the likelihood of not developing hypotension after intrathecal injection.
- Levobupivacaine (LB) 12 mg (Placebo Comparator): Patients will be stratified into three groups by 80 patients: those who will receive 6, 8 or 12 mg of Levobupivacaine intrathecally (Chirocaine, Abbot Laboratories, amp. 5 mg/ml). Patients will receive 12 mg of Levobupivacaine alone intrathecally.
  Hemodynamic side effects will be recorded after intrathecal injection. The level and duration of sensory block, time until two-segment regression, T12 regression andl full skin sensory sensibility at the S1 segment will be registered
  Interventions: Drug: The impact of 10 independent variables on the likelihood of not developing hypotension after intrathecal injection.

INTERVENTIONS:
Drug: The impact of 10 independent variables on the likelihood of not developing hypotension after intrathecal injection. — The study will be conducted to assess the impact of a 10 independent variables (dose and combination of Levobupivacaine with Fentanyl or Sufentanil, age, basal systolic blood pressure (SBP), basal mean arterial pressure (MAP), time to lowest spinal SBP, upper limit of sensory block (dermatoma level), time intervals of sensory recovery for two consecutive dermatoma level (two-segment regression), time intervals of sensory recovery to the twelfth thoracic dermatoma (T12 regression), time intervals of sensory recovery to the first sacral dermatoma (S1 regression) and Body Mass Index) on the likelihood of not developing hypotension after intrathecal injection.
  Other Names: levobupivacaine

SUMMARY:
To find the optimal dose and combination of small dose of Levobupivacaine (LB) coadministered intrathecally with Fentanyl (F) or Sufentanil (S) with the highest probability for not developing hypotension and the lowest opioid side effect that would be sufficient to achieve and maintain a sensory block to the tenth thoracic dermatoma (T10) in elderly patients for surgery lasting > 45 minutes as compared with large dose of Levobupivacaine alone.

DETAILED DESCRIPTION:
Hypotension and bradycardia are the most common adverse hemodynamic effects associated with spinal anesthesia, with particular frequency among the elderly. These complications are more hazardous in the elderly because they may have decreased physiological reserves and compromised blood supply to various vital organs. Hypotension is mainly related to the spinal anesthesia block height. One approach to improve hemodynamic stability is to use smaller doses of local anesthetic (< 10 mg of Levobupivacaine) to limit the distribution of local anesthetic within the subarachnoid space and hence to limit the block height. However, a smaller dose of local anesthetic may increase the incidence of inadequate level of sensory anesthesia for the anticipated surgery as compared with larger doses (> 10 mg of Levobupivacaine). Another concern about smaller dose of local anesthetic is the inadequate duration of sensory anesthesia. Therefore, small dose of local anesthetic need to be combined with opioids (Fentanyl or Sufentanil). However, intrathecal opioids are associated with several side effects such as pruritis, nausea, vomiting, shivering and respiratory depression. This will be the first comparative study of two small doses of Levobupivacaine (6 and 8 mg) combined using intrathecal Fentanyl (F, 25 and 35 mcg) or Sufentanil (S, 5 and 7 mcg) compared with large dose of Levobupivacaine alone (12 mg) in spinal anesthesia. The study will be conducted to assess the impact of a 10 independent variables (dose and combination of Levobupivacaine with Fentanyl or Sufentanil, age, basal systolic blood pressure (SBP), basal mean arterial pressure (MAP), time to lowest spinal SBP, upper limit of sensory block (dermatome level), time intervals of sensory recovery for two consecutive dermatome level (two-segment regression), time intervals of sensory recovery to the twelfth thoracic dermatoma (T12 regression), time intervals of sensory recovery to the first sacral dermatoma (S1 regression) and Body Mass Index) on the likelihood of not developing hypotension after intrathecal injection. The goal of the study is to find an optimal dose and combination of Levobupivacaine and Fentanyl or Sufentanil with the highest probability of not developing the hypotension as well as with the lowest opioid side effect that would be potent enough in achieving and maintaining a sensory block at T10 level for surgery lasting more than 45 minutes in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* male patients
* ASA II-III undergoing elective urological (transuretheral or transvesical prostatectomy, hydrocelectomy, orchiectomy) or lower abdominal (inguinal herniorrhaphy) surgery under spinal anesthesia requiring a sensory block to at least the tenth thoracic dermatoma, lasting >45 minutes.

Exclusion Criteria:

* severe systemic disorders
* patients unwilling to accept regional anesthesia
* patients who will develope sensory block level lower than T10 dermatoma after intrathecal injection
* patients with an abnormal coagulation profile or with significant pulmonary disease (reactive airway disease or chronic obstructive pulmonary disease requiring daily bronchodilator or steroid use and/or room air oxygen saturation <95% immediately before surgery).

Ages: 65 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Optimal dose and combination of Levobupivacaine and Fentanyl or Sufentanil in elderly patients | 9 months
  To find an optimal dose and combination of Levobupivacaine and Fentanyl or Sufentanil with the highest probability of not developing the hypotension as well as with the lowest opioid side effect that would be potent enough in achieving and maintaining a sensory block at T10 level for surgery lasting more than 45 minutes in elderly patients. Binary logistic regression will be performed to assess the impact of a number of factors on the likelihood that patients may not develop hypotension. The model will consists of 10 independent variables (dose and combination of levobupivacaine with Fentanyl or Sufentanil, age, basal SBP, basal MAP, time to lowest spinal SBP, upper limit of sensory block, time until two-segment regression, time until T12 regression, time until S1 regression, BMI).

CONTACTS AND LOCATIONS:
Overall Officials: Jadranka Pavičić Šarić, PhD, Principal Investigator — University Hospital Merkur
Locations (1):
- University Hospital Merkur, Zagreb, Croatia, Croatia